CLINICAL TRIAL: NCT05107648
Title: Gardner GOALS for Treatment of Obesity
Brief Title: Gardner Packard Healthy Lifestyles Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Elizabeth Shepard, Clinical Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53309
Record Dates: First submitted 2021-10-20; First posted 2021-11-04 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gardner GOALS (Experimental): Healthy lifestyle intervention by telehealth plus regular clinic visits
  Interventions: Behavioral: Gardner GOALS
- Control (No Intervention): Regular clinic visits

INTERVENTIONS:
Behavioral: Gardner GOALS — 12 lesson curriculum focusing on healthy eating, increased physical activity and decreased screen time
  Arms: Gardner GOALS

SUMMARY:
Gardner GOALS is a 6 month program for treatment of childhood obesity that consists of twice monthly telehealth meetings with a health educator. Potential participants enter the study using a randomly ordered list of eligible patients based on BMI, age and number of clinic visits in 2020.

DETAILED DESCRIPTION:
The Gardner GOALS curriculum focuses on healthy eating and activity. The study participants are kids 6 to 14 years old with BMI ≥95th percentile who are patients at the Gardner Packard Children's Health Center, a federally qualified health center. Lessons contain educational materials and behavioral change strategies to promote healthy eating and physical activity and reduce screen time. Patients are encouraged to continue routine clinic visits with their primary care physicians during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 95th percentile
* Two clinic visits in 2020

Exclusion Criteria:

* Signs of an eating disorder
* Moved out of town and not planning to return to Gardner Packard Children's Health Center

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Body mass index | Baseline, year 1
  Change in trajectory of body mass index from the year prior to the intervention compared to the year after starting the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shepard, MD, Study Director — Stanford University
Locations (1):
- Gardner Packard Children's Health Center, Atherton, California, United States

IPD SHARING:
Plan to Share IPD: No